CLINICAL TRIAL: NCT02317328
Title: Adaptive Optics Retinal Imaging
Status: Recruiting | Type: Observational
Sponsor: National Eye Institute (NEI) (NIH)
Responsible Party: Sponsor
Organization: National Institutes of Health Clinical Center (CC) (NIH)
Other Study IDs: 150020; 15-EI-0020
Record Dates: First submitted 2014-12-13; First posted 2014-12-16 (Estimated); Last update posted 2026-01-28 (Actual); Status verified 2026-01-23

CONDITIONS: Eye Diseases; Healthy Volunteers
Keywords: Eye Disease; Natural History
MeSH Terms: conditions — Eye Diseases

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Cross-Sectional
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Affected participants: Participants with ocular conditions
- Healthy Volunteers: Healthy volunteers

SUMMARY:
Background:

- By the time diseases of the retina are detected, serious damage has often already been done. Researchers want to find better ways of viewing the retina. One way called adaptive optics may help detect problems earlier.

Objectives:

- To study if adaptive optics can help find better ways to diagnose, treat, and manage retinal diseases.

Eligibility:

* People over age 12 with an eye disease.
* Healthy volunteers over age 12.

Design:

* Participants will be screened with medical history and eye exams. These may include dilating pupils and taking pictures of the eyes.
* Participants will have 1 or more study visits. They will have:
* Medical and eye history.
* Questions about their medications.
* Eye exam including pupil dilation.
* Adaptive optics imaging. After dilation, participants sit still while looking into an adaptive optics instrument. They look at specific places and images are taken of their retina.
* They may also have:
* More images.
* Perimetry. Participants look into a lens and press a button when they see a light.
* Color vision tests.
* Electroretinogram. Participants will get numbing eye drops and special contact lenses. A small metal electrode will be put on their forehead. They will look at flashing lights and try not to blink.

DETAILED DESCRIPTION:
Objective: The objective of this protocol is to collect and assess adaptive optics (AO) retinal images of normal and diseased eyes.

Study Population: Three hundred and fifty (350) participants with eye diseases and 250 normal volunteers will be enrolled.

Design: This is an observational protocol which will enroll 350 participants with various eye diseases and 250 age-matched healthy volunteers over five years. In general, participants will undergo a complete ophthalmic examination including assessments of visual acuity, intraocular pressure, and a dilated ocular examination. Imaging will be performed using adaptive optics instruments deployed in the NEI Eye Clinic.

Outcome Measures: The primary outcome for this protocol is qualitative and quantitative assessment of the AO images with comparisons of normal and diseased states.

ELIGIBILITY:
* INCLUSION CRITERIA:

Participants will be eligible if they:

* Are 12 years of age or older.
* Have the ability to cooperate with an eye exam and adaptive optics imaging.
* Have the ability to understand and sign an informed consent or have a parent/legal guardian to do so if they are minor children.
* Have an eye disease or are a healthy volunteer with a normal eye exam (no visually-significant eye findings on examination).

EXCLUSION CRITERIA:

Participants will not be eligible if:

-They have a condition which prevents adequate images from being obtained (e.g. unstable fixation or media opacity).

EXCLUSION CRITERIA FOR FLUORESCEIN AND/OR INDOCYANINE GREEN IMAGING

Partaicipants are not eligible for fluorescein and/or indocyanine green imaging if they:

* Are under 18 years of age.
* For participants who will undergo fluorescein imaging have a history of adverse reaction to fluorescein.
* For participants who will undergo indocyanine green imaging have a history of adverse reaction to indocyanine green dye, know or suspected allergies to iodine or shellfish.

Ages: 12 Years to 120 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Study Population: 500 participants with eye diseases and 500 healthy volunteers will be enrolled.
Sampling Method: Non-Probability Sample
Enrollment: 1000 (Estimated)
Dates: Start 2015-02-20 (Actual); Primary Completion 2028-03-31 (Estimated); Study Completion 2028-03-31 (Estimated)

PRIMARY OUTCOMES:
Qualitative and quantitative assessment of AO images | ongoing
  Qualitative and quantitative assessment of AO images with comparison of normal and diseased states.

CONTACTS AND LOCATIONS:
Overall Officials: Johnny C Tam, Ph.D., Principal Investigator — National Eye Institute (NEI)
Locations (1):
- National Institutes of Health Clinical Center, Bethesda, Maryland, United States

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Background] Hendrickson A, Drucker D. The development of parafoveal and mid-peripheral human retina. Behav Brain Res. 1992 Jul 31;49(1):21-31. doi: 10.1016/s0166-4328(05)80191-3. PMID 1388798
- [Background] Wing GL, Blanchard GC, Weiter JJ. The topography and age relationship of lipofuscin concentration in the retinal pigment epithelium. Invest Ophthalmol Vis Sci. 1978 Jul;17(7):601-7. PMID 669891
- [Background] Fotedar R, Wang JJ, Burlutsky G, Morgan IG, Rose K, Wong TY, Mitchell P. Distribution of axial length and ocular biometry measured using partial coherence laser interferometry (IOL Master) in an older white population. Ophthalmology. 2010 Mar;117(3):417-23. doi: 10.1016/j.ophtha.2009.07.028. Epub 2010 Jan 19. PMID 20031227
- See also: NIH Clinical Center Detailed Web Page — https://clinicalstudies.info.nih.gov/cgi/detail.cgi?A_2015-EI-0020.html